CLINICAL TRIAL: NCT00580853
Title: The Effect of Varenicline (Chantix) and Bupropion (Zyban) on Smoking Lapse Behavior
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0702002390; P50AA015632 (NIH)
Record Dates: First submitted 2007-12-25; First posted 2007-12-27 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-01

CONDITIONS: Smoking Lapse Behavior
Keywords: smoking lapse behavior; smoking cessation; varenicline; bupropion; medication effect on smoking lapse behavior
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline; Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- varenicline (Experimental): varenicline 2mg/day
  Interventions: Drug: varenicline
- Bupropion (Experimental): Bupropion 300mg/day
  Interventions: Drug: bupropion
- Placebo (Placebo Comparator): Placebo Control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: varenicline — 2mg/day, with 1-week lead-in medication period The starting dose is 0.5 mg/day for days 1-2, followed by 0.5mg twice daily for days 3-5 and then 1mg twice daily for days 4-7. 1mg administered during laboratory session (day 8).
  Other Names: Chantix
  Arms: varenicline
Drug: bupropion — 300mg/day, with 1-week lead-in medication period The starting dose is 150mg/day for days 1-3, 300mg/day for days 4-7. 300mg administered during laboratory session (day 8).
  Other Names: Zyban
  Arms: Bupropion
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine how smoking cessation medications (varenicline, bupropion) affect the ability to resist smoking and also subsequent ad-lib smoking in non-treatment seeking daily smokers.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-55
* able to read and write in English
* Smokers

Exclusion Criteria:

* any significant current medical or psychiatric conditions that would contraindicate smoking
* current Diagnostic and Statistical Manual IV abuse or dependence of other substances, other than nicotine dependence or alcohol abuse
* positive test result at intake appointments on urine drug screens conducted for opiates, cocaine, or benzodiazepines
* women who are pregnant or nursing
* suicidal, homicidal, or evidence of current severe mental illness
* participants prescribed any psychotropic drug in the 30 days prior to study enrollment
* blood donation within the past 6 weeks
* individuals seeking treatment for smoking cessation or have attempted to quit smoking within the past 3 months
* specific exclusions for bupropion administration not already specified, including: have taken monoamine inhibitors in the past 6 weeks; history of anorexia or bulimia; previous hypersensitivity to bupropion; history of alcohol or drug dependence in the past year; history of seizure disorder of any etiology
* known allergy to varenicline or taking H2blockers
* participation within the past 8 weeks in other studies that involve additive blood sampling and/or interventional measures that would be considered excessive in combination with the current study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2007-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation, Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Bupropion | Placebo
Started | 20 | 21 | 21
Completed | 20 | 21 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Bupropion | Placebo | Total
Number analyzed (Participants) | 20 | 21 | 21 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.95 (11.36) | 34.95 (9.70) | 36.47 (10.95) | 35.47 (6.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 9 | 26
  Male | 11 | 13 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Latency to Initiate Ad-lib Smoking Session
Description: minutes to start smoking (range 0 to 50 minutes)
Time Frame: 0 to 50 minutes
Population: Subsample with high nicotine dependence
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Varenicline | Bupropion | Placebo
Number analyzed (Participants) | 8 | 9 | 10
minutes | 38.138 (6.268) | 39.416 (5.939) | 19.249 (6.196)

2. Secondary Outcome: Number of Cigarettes Smoked During the 60 Minute Ad-lib Period
Description: number of cigarettes smoked (range 0-8) during the 60 minute ad-lib period
Time Frame: 60 minutes
Measure: Mean (Standard Error); unit: number of cigarettes
Arm/Group | Varenicline | Bupropion | Placebo
Number analyzed (Participants) | 20 | 21 | 21
number of cigarettes | .713 (.351) | 1.287 (.342) | 2.085 (.396)

ADVERSE EVENTS:
Time Frame: Titration period (7 days)
Description: All adverse events reported during 1 week medication period. Baseline reporting not controlled. Subjects were queried about the presence/absence of severity of common symptoms (>5% from placebo according to manufacturer) associated with varenicline and bupropion. Adverse events assessed on Day 2 and Day 8.
Arm/Group | Varenicline | Bupropion | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 13/20 | 13/21 | 13/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=20) | Bupropion (N=21) | Placebo (N=21)
Nausea (Gastrointestinal disorders) | 3 | 3 | 0
need to urinate (Renal and urinary disorders) | 5 | 3 | 2
Dry mouth (General disorders) | 2 | 2 | 2
Insomnia (General disorders) | 2 | 2 | 1
Flatulence (Gastrointestinal disorders) | 3 | 4 | 3
Abnormal dreams (General disorders) | 3 | 1 | 1
Discomfort (General disorders) | 0 | 2 | 1
Headache (General disorders) | 2 | 3 | 4
Change in taste (General disorders) | 2 | 4 | 2
Runny nose (General disorders) | 6 | 2 | 3
Change in appetite (General disorders) | 2 | 4 | 4
Trouble concentrating (General disorders) | 2 | 2 | 2
Sweating (General disorders) | 0 | 4 | 1
Heartburn (Gastrointestinal disorders) | 2 | 2 | 1
Cough (General disorders) | 1 | 1 | 2
Drowsiness (General disorders) | 2 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No